CLINICAL TRIAL: NCT06783231
Title: Implications of Identification With the Aggressor (IWA) : a Randomized Control Trial
Brief Title: Identification With the Aggressor (IWA)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, Yael Lahav, Prof. Yael Lahav, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0009390-2
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Female; Abuse Neglect; Abuse Physical; Abuse, Child
Keywords: identification with the aggressor; abuse; trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial comprising of 2 assessments :before (T1) and after (T2) experimental manipulation. Participants with and without history of interpersonal abuse will be randomly allocated to one of three study conditions and will receive different instructions before listening to the audio recording of the identification with the aggressor (IWA) lab task: (1) The 'identification with the aggressor' group will be asked to try to identify, understand and adopt the point of view of the perpetrator; (2) The 'identification with the victim' group will be asked to try to identify, understand and adopt the point of view of with the victim; (3) The control group will be asked to pay attention to the story's details and to try and remember as much details as they can.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The 'identification with the aggressor' group (Experimental): In this experimental group participants will be asked to try to identify, understand and adopt the point of view of Lori (the perpetrator), before listening to the audio recording portraying a romantic relationship between two women (Lori and Sophia), in which one of them (Lori - the perpetrator) is being aggressive towards the other (Sophia - the victim).
  Interventions: Behavioral: Identifying with the aggressor
- The 'identification with the victim' group (Active Comparator): In this experimental group participants will be asked to try to identify, understand and adopt the point of view Sophia (the victim), before listening to the audio recording portraying a romantic relationship between two women (Lori and Sophia), in which one of them (Lori - the perpetrator) is being aggressive towards the other (Sophia - the victim).
  Interventions: Behavioral: Identifying with the victim
- The control group (Placebo Comparator): In this experimental group participants will be asked to pay attention to the story's details and to try and remember as much details as they can, before listening to the audio recording portraying a romantic relationship between two women (Lori and Sophia), in which one of them (Lori - the perpetrator) is being aggressive towards the other (Sophia - the victim).
  Interventions: Behavioral: Neutral

INTERVENTIONS:
Behavioral: Identifying with the aggressor — The IWA lab task consists 10 min audio recorded story, portraying a romantic relationship between two women (Lori and Sophia), in which one of them (Lori - the perpetrator) is being aggressive towards the other (Sophia - the victim). The story was carefully designed to align with ethical considerations - it is non-graphic, contains no severe acts of violence, and mostly describes a romantic power dynamic which may be considered abusive or toxic. The three groups of participants will receive different instructions before listening to the audio recording. The 'identification with the aggressor' group will be asked to try to identify, understand and adopt the point of view of Lori (the perpetrator)
  Arms: The 'identification with the aggressor' group
Behavioral: Identifying with the victim — The IWA lab task consists 10 min audio recorded story, portraying a romantic relationship between two women (Lori and Sophia), in which one of them (Lori - the perpetrator) is being aggressive towards the other (Sophia - the victim). The story was carefully designed to align with ethical considerations - it is non-graphic, contains no severe acts of violence, and mostly describes a romantic power dynamic which may be considered abusive or toxic. The three groups of participants will receive different instructions before listening to the audio recording. The 'identification with the victim' group will be asked to try to identify, understand and adopt the point of view of Sophia (the victim)
  Arms: The 'identification with the victim' group
Behavioral: Neutral — The IWA lab task consists 10 min audio recorded story, portraying a romantic relationship between two women (Lori and Sophia), in which one of them (Lori - the perpetrator) is being aggressive towards the other (Sophia - the victim). The story was carefully designed to align with ethical considerations - it is non-graphic, contains no severe acts of violence, and mostly describes a romantic power dynamic which may be considered abusive or toxic. The three groups of participants will receive different instructions before listening to the audio recording. The control group will be asked to pay attention to the story's details and to try and remember as much details as they can.
  Arms: The control group

SUMMARY:
This is a randomized control study, comprising of 2 assessments :before (T1) and after (T2) the identification with the aggressor (IWA) lab task.

DETAILED DESCRIPTION:
Background: Abuse is a severe trauma that has multiple psychological implications. One of the most paradoxical effects of CA is the identification with the aggressor (IWA) phenomenon. Research to date has indicated associations between IWA and various negative outcomes, such as PTSD, dissociation, guilt, suicidality, and increased likelihood of returning to abusive relationships . Nonetheless, these studies were based on a cross-sectional design, and thus excluded the possibility of establishing causality or shedding light on the complex dynamics of IWA. In addition, to the best of our knowledge, no experimental research has been conducted on IWA thus far. This type of study is required to examine causal relationships between IWA and potential outcomes. In an attempt to bridge this gap, the current study will serve as a pilot study examining the efficacy of a new lab task designed to ethically but validly manipulate a state of IWA among women with and without a history of abuse. Developing a tool that experimentally manipulates IWA under laboratory conditions will allow examining the influences of IWA, while controlling for other consequences of the abuse, trauma, or life circumstances. In order to test the effectiveness of our lab task, the investigators will compare measurements of relevant outcomes before and after the task in the process.

Methods:

This is a randomized controlled trial comprising of 2 assessments :before (T1) and after (T2) experimental manipulation. Participants with and without history of interpersonal abuse will be randomly allocated to one of three study conditions and will receive different instructions before listening to the audio recording of the identification with the aggressor (IWA) lab task: (1) The 'identification with the aggressor' group will be asked to try to identify, understand and adopt the point of view of the perpetrator; (2) The 'identification with the victim' group will be asked to try to identify, understand and adopt the point of view of with the victim; (3) The control group will be asked to pay attention to the story's details and to try and remember as much details as they can.

Population: the investigators will recruit 300 female adults with and without history of interpersonal abuse. Participants with a history of interpersonal abuse will be identified via questionnaires during screening. The sample size was calculated based on power analyses via G*Power 3 software derived from p-value of .05 and statistical power of .80.

Tools: outcome measures will be consist self-report questionnaires as well as Reading the Mind in the Eye Test (RMET; Baron-Cohen et al., 2001) and two new versions of Implicit Association Tests (IAT; Greenwald, McGhee & Schwartz, 1998) created for the purpose of the present study. The experimental manipulation will comprise of the identification with the aggressor (IWA) lab task.

Expected Results: Findings may advance the understanding both mechanisms at the basis of IWA as well as its effects, and in this way may contribute to developing preventative measures for IWA among abuse survivors.

ELIGIBILITY:
Inclusion Criteria:

* Good command of Hebrew language
* Age 18 or older

Exclusion Criteria:

* Diagnosis of dissociative identity disorder
* Persistent drug use
* Diagnosis of autism spectrum disorder.
* Hearing or vision difficulties (that may impair the experimental manipulation and participants' ability to complete the Reading the Mind in the Eyes and the IAT tasks).
* Being currently subjected to abuse
* Suicidal risk, as assessed by a clinical interview.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals who identify themselves as women
Enrollment: 300 (Estimated)
Dates: Start 2003-04-02 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
International Trauma Questionnaire (ITQ) | Change between T1 and T2: (48 hours before and immediately after the manipulation= The IWA lab task)
  The ITQ is an 18-items self-report measure focusing on the core features of Complex PTSD and PTSD. This questionnaire was developed to be consistent with the organizing principles of the ICD-11. The current literature suggests that the ITQ is a valid tool for the assessment of ICD-11 PTSD and CPTSD, with good psychometric properties.
PTSD Checklist for DSM-5 (PCL-5) | Change between T1 and T2: (48 hours before and immediately after the manipulation= The IWA lab task)
  The PCL-5 is a 20-item self-report questionnaire that examines the presence of the 20 PTSD symptoms listed in the DSM-5. The PCL-5 has a variety of purposes including screening individuals for PTSD and making a provisional PTSD diagnosis. The recommended cut-off for the assessment of PTSD using this tool is 33. The PCL-5 is a very reliable and valid assessment tool for PTSD, with abundant literature that supports its excellent psychometric properties.
Patient Health Questionnaire-9 (PHQ-9) | Change between T1 and T2: (48 hours before and immediately after the manipulation= The IWA lab task)
  A modified version of the nine-item Patient Health Questionnaire-9 will be used to assess depression symptoms. Participants will rate the frequency (from 0 - not at all, to 3 - nearly every day) in which they were bothered by each depression symptom in the last two weeks. Total PHQ-9 score will be created by summing ratings for all symptoms.
Identification with the Aggressor Scale (IAS) | Change between T1 and T2: (48 hours before and immediately after the manipulation= The IWA lab task)
  Levels of IWA will assess via IAS, a 23-item self-report questionnaire. The items will be presented to the participants as reflecting "possible reactions that people may experience as a result of abuse or offense". Participants will be asked to rate on an 11-point Likert scale, ranging from 0% (never) to 100% (all the time), the frequency with which they experienced each manifestation of IWA. The scale comprises four subscales: adopting the perpetrator's experience concerning the abuse ; identifying with the perpetrator's aggression ; replacing one's agency with the perpetrator's ; and becoming hypersensitive to the perpetrator . The IAS has
The Interpersonal Trauma Doubt Scale (ITDS) | Change between T1 and T2: (48 hours before and immediately after the manipulation= The IWA lab task)
  Doubt regarding judgments and assessments about the characteristics of the abuse will be assessed via The Interpersonal Trauma Doubt Scale (ITDS). This questionnaire comprises of 10 items tapping one's doubts concerning judgments regarding oneself, the perpetrator, and the abuse.
Difficulties in Emotion Regulation Scale (DERS-18) | Change between T1 and T2: (48 hours before and immediately after the manipulation= The IWA lab task)
  A short form of the DERS is a self-report scale consists of 18-Items, rated on a 5-point scale that measures emotion regulation in the following subscales: 1. Nonacceptance of emotional responses 2. Difficulty engaging in goal-directed behavior 3. Impulse control difficulties 4. Lack of emotional awareness 5. Limited access to emotion regulation strategies 6. Lack of emotional clarity. The DERS has good internal consistency and good test-retest reliability.
Maudsley Violence Questionnaire (MVQ) | Change between T1 and T2: (48 hours before and immediately after the manipulation= The IWA lab task)
  The MVQ is a 54-item questionnaire covering a range of cognitions (beliefs, rules, distortions and attributions) that may provide support, justifications or injunctions to violence. Each item is rated on a 5-point Likert scale, ranging from 1 to 5. The MVQ comprises two subscales: 1) Machismo (42 items) relates to embarrassment over backing down, justification of violence in response to threat and attack, violence as part of being male and strong and the weakness associated with fear and non-violence; 2) Acceptance of violence (14 items) including overt enjoyment and acceptance of violence (in the media and in sport) and injunctions against or rejection of violence as an acceptable behaviour. For the purpose of the study only the Acceptance of violence subscale will be utilized.
Reading the Mind in the Eye Test (RMET) | T2: (immediately after the manipulation= The IWA lab task)
  RMET is a social cognition measure that examines a participant's ability to identify complex emotions and mental states. Participants will be presented with 36 images of human eyes and will be asked to choose out of 4 words the one that best describes the emotion the person in the image is experiencing. Social cognition will be measured by the number of overall correct answers in the task as well as the response time for correct answers.
Implicit Association Test (IAT) - new version attitudes towards the characters of the IWA task | T2: (immediately after the manipulation= The IWA lab task)
  The IAT is a computerized screening test developed by Greenwald and is designed to examine hidden attitudes. A new version was created for the purpose of the current study to examine attitudes towards the characters which are part of the IWA task (Lori, the perpetrator and Sophia the victim. These attitudes will be assessed by measuring automatic links between the characters (for example "Lori" versus "Sophia ") and attributions ("good" or "bad"). The test has seven stages in which the participants are required to classify words into different categories as quickly as possible By pressing the right ("k")/left ("D") key, the reaction time and the number of errors in the cross-category steps will reflect the strength of the implicit beliefs about the characters which are part of the IWA task.
Implicit Association Test (IAT) - new version attitudes regarding harm/violent behavior | T2: (immediately after the manipulation= The IWA lab task)
  The IAT is a computerized screening test developed by Greenwald and is designed to examine hidden attitudes. A new version was created for the purpose of the current study to examine attitudes towards the legitimacy of harm/violent behavior. These attitudes will be assessed by measuring automatic links between certain concepts (for example "abuse" versus "love") and attributions (for example "permitted" or "forbidden"). The test has seven stages in which the participants are required to classify words into different categories as quickly as possible By pressing the right ("D")/left ("K") key, the reaction time and the number of errors in the cross-category steps will reflect the strength of the implicit beliefs regarding the legitimacy of harm/violent behavior.
Dissociative Experiences Scale-II (DES-II) | Change between T1 and T2: (48 hours before and immediately after the manipulation= The IWA lab task)
  Dissociation will be measured by the DES-II, a 28-item self-report questionnaire that measures the frequency of dissociative experiences. The total dissociative score is computed as the mean of items, ranging from 0 to 100. The DES-II has been shown to have high validity and reliability.
The Selflessness scale (SS) | Change between T1 and T2: (48 hours before and immediately after the manipulation= The IWA lab task)
  The SS is a 15-item questionnaire on a four-point Likert scale that measured altruism by quantifying the tendency to ignore one's own needs and interests and serve the needs of others. The items ask about sacrifice for family and others, self-denial, and lack of self-interest.
7. Sense of Body Boundaries Survey (BBS) | T2: (immediately after the manipulation= The IWA lab task)
  A subjective feeling of a disturbance or disruption of the body's boundaries will assess via 17 items self-report questionnaire, divided into two scales: one refers to the subject's sense of physical separation from his environment and is called "The barrier subscale" (for example: "I do not feel tangibly separated from the reality surrounding me"), the second is a permeability scale (known as: "The permeability subscale"), and refers to the feeling of physical vulnerability (for example: "Sometimes I imagine/experience my body as a wide open window"). Subjects will be asked to answer on a scale of 1-5, according to their degree of identification with the physical sensation or physical experience presented in the item.

SECONDARY OUTCOMES:
Manipulation check questions | T2: (immediately after the manipulation= The IWA lab task)
  To make sure that the task was indeed understood as intended and evoked the desired emotions and cognitions participants will be asked to answer 25 Manipulation check questions (e.g., "How much did you relate to the character of Lori?"; "To what extent did you experience a change in your ability to understand Lori's point of view?")
The short form of the Childhood Trauma Questionnaire (CTQ-SF) | Baseline ( screening phase)
  Participants with a history of interpersonal abuse will be identified via the CTQ-SF. For the purpose of this study, only 15 items referring to emotional, physical, or sexual abuse were utilized. Based on previous research, participants were classified as having a history of childhood abuse if they scored above any of the following cut-off scores: for physical abuse (>8), sexual abuse (>6), and emotional abuse (>9).
Characteristics of the assault | Baseline ( screening phase)
  The characteristics of the continuous assault will be examined using a questionnaire that was designed for the purpose of this study. Participants will be asked to indicate which assault they have experienced by marking from an existing list with an open option of adding additional events. The questionnaire also includes additional questions about the characteristics of the assault, such as at what age it occurred, how long it lasted, and questions about the nature of the relationship with the perpetrator. Further questions will refer to the behavior of the perpetrator and the reaction of the participant at the time of the assault.
Open questions | T2: (immediately after the manipulation= The IWA lab task)
  We will ask participants 3 Open questions on their experience during the manipulation: 1) What did you feel while listening to the audio recorded story? 2) How do you feel about Lori? 3) 2. How do you feel about Sophia?
Background questionnaire | Baseline ( screening phase)
  A brief demographic questionnaire that assessed gender, age, education, and relational status. The questionnaire will also include questions about treatment, such as whether the participant is currently receiving psychological or psychopharmacological treatment, the type of treatment or medication, and whether they have received a psychiatric diagnosis. Additionally, participants will be asked to describe the chronic traumatic event they have experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Yael Lahav, Phd, Principal Investigator — Tel Aviv University; Danny Horesh, Phd, Principal Investigator — Bar Ilan University

IPD SHARING:
Plan to Share IPD: No
Due to the nature of this research, participants of this study did not agree for their data to be shared publicly, so supporting data is not available.